CLINICAL TRIAL: NCT03047200
Title: Pancreatic Islet Cell Transplantation After Kidney Transplantation - A Novel Approach to Immunosupression
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: There were not patients that meet inclusion/exclusion criteria. Site decided to close study.
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 008-189
Record Dates: First submitted 2016-05-04; First posted 2017-02-08 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Islet Cell Transplantation; Type 1 Diabetes
Keywords: Diabetes Mellitus; Hypoglycemia; Hyperglycemia; Type 1 Diabetes; Islet Cell Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hypoglycemia; Hyperglycemia | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Islet cell transplantation — The process is based on the enzymatic isolation of the pancreatic islets of Langerhans from an organ procured from a cadaveric donor; the islets obtained are injected into the liver of the recipient via percutaneous catheterization of the portal venous system . This procedure allows the selective transplantation of the insulin-producing cell population avoiding open surgery as well as the transplantation of the duodenum and the exocrine pancreas and their related morbidity.

SUMMARY:
The purpose of this study is to further test islet cell transplant in patients who have had a kidney transplant. This study will also evaluate the safety and effectiveness of the anti-rejection medications used to prevent rejection after your islet cell transplant.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) type 1 is a disease with significant social and economic impact. The prevalence of the disease in the United States is about 120,000 in individuals aged 19 or less and 300,000 to 500,000 at all ages and 150 million worldwide. There are 30,000 new cases diagnosed each year in the United States. DM is one of the most frequent chronic diseases in children in the United States 1. The cost of treatment and complications of this disease in the United States is 90 billion dollars a year.

To date there are no mechanical devices able to effectively adjust the dose of insulin injected according to the serum glucose levels in patients with DM. This leads to less-than-perfect sugar control, with episodes of hypoglycemia which can be dangerous.

The emerging alternative to whole organ pancreas transplantation is pancreatic islet cell transplantation (ICT). The process is based on the enzymatic isolation of the pancreatic islets of Langerhans from an organ procured from a cadaveric donor 13-15; the islets obtained are injected into the liver of the recipient via percutaneous catheterization of the portal venous system 16. This procedure allows the selective transplantation of the insulin-producing cell population avoiding open surgery as well as the transplantation of the duodenum and the exocrine pancreas and their related morbidity.

The initial efforts with ICT had only modest results. The immunosuppression regimen was similar to the one used in solid organ transplantation, based on high dose steroids and calcineurin inhibitors - both agents with diabetogenic effects. The results improved markedly with the changes in the manipulations of the islets, and the change in immunosuppression thus avoiding the higher doses of steroids and using sirolimus, tacrolimus and daclizumab initiated by the investigators group at the University of Alberta in Edmonton, Canada. Their protocol requires in general two islet cell infusions in order to attain the critical cell mass necessary to achieve insulin-independency. The changes in treatment were adopted as the Edmonton Protocol, which is used in several transplant centers, worldwide.

Isolation of the islets from donor pancreata will occur in the Baylor University Medical Center Islet Cell Processing Laboratory (ICPL). The islet cell infusion is performed in the Interventional Radiology Suite at Baylor University Medical Center or Baylor All Saints Medical Center by an interventional radiologist. The procedure takes place in a suite designed for invasive procedures using sterile technique with access to general anesthesia if necessary. Following the procedure the patient is observed in the Interventional Radiology recovery area for as long as necessary as determined by a Physician and then transferred to the Transplant Service for an overnight stay. After recovery, the patient is admitted to the hospital on the Transplant Service for a 1-2 day observation.

The focus of the research in the ICT is centered on the development of a safe and effective procedure that will eventually replace surgical pancreas transplantation together with an ideal immunosuppressive regimen that provides safe and effective prevention against rejection, while minimizing the adverse events associated that negatively impact transplant recipient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been fully informed and has signed an IRB approved informed consent form and is willing and able to follow study procedures for the full 24 months.
2. Type 1 diabetes mellitus of more than 5 years duration
3. Age between 18 and 65
4. Unstable diabetes mellitus control despite expert management by a diabetology care team for at least 6 months prior to consideration for transplantation as defined by the following:

   * During the past six months (or during the period of intensive diabetes care): Any episodes of hypoglycemic unawareness, as defined by the inability to recognize glucose levels below 50 mg/dL; or episodes of loss of cognitive function; or frequent episodes of symptomatic hypoglycemia; or admission to the hospital for hypo- or hyperglycemia; and
   * HbA1C>6.5%.
5. Patient underwent kidney transplantation at least six months before enrollment, and has stable kidney allograft function, defined as creatinine levels of maximum 2 mg/dl, stable renal allograft function as assessed by the transplant nephrologist, and has a creatinine clearance of more than 40 ml/min.
6. Psychogenically able to comply, in the opinion of the investigator
7. Female patients of childbearing potential must have a negative urine or serum pregnancy test upon hospitalization or within 7 days prior to enrollment and have agreed to utilize effective birth control throughout the study as well as for 6 weeks following study completion

Exclusion Criteria:

* Patient has previously received or is receiving an organ or bone marrow transplant other than a first kidney transplant.

  2. Patient has a known hypersensitivity to Tacrolimus, Sirolimus, Alemtuzumab, or Mycophenolate (allow substitution of Myfortic for CellCept).

  3. Patient is pregnant or lactating (must provide effective contraception method).

  4. Patient has participated in a blinded trial or participated in a trial involving a non-marketed (investigational) drug within 3 months of enrollment.

  5. Patient has participated in a trial involving a marketed drug or an infusion device within 30 days of the start of the trial.

  6. Patient exhibits any one of the following clinical criteria:
  * Creatinine clearance or Glofil test < 40 mL/min
  * Serum creatinine > 2.0 mg/dL consistently, or more than 0.2 mg/dl increase in creatinine over the last five months
  * Body mass index > 28
  * Malignancy other than BCC and SCC
  * Radiographic evidence of pulmonary infection
  * Evidence of liver disease as evidenced by >2X ULN for AST, ALT, Alk. Phos., or T. bili.
  * Active infections
  * Hypercoagulable states (history of recurrent venous thrombosis, defined thrombophilia)
  * Bleeding / coagulation disorders
  * Basal C-peptide > 0.3 ng/mL
  * HbA1C >12%
  * Insulin requirement > 1 IU/kg/day
  * Seropositivity for HIV, HBV, HCV, HTLV-I
  * Abnormal Pap smear, active gynecological infection
  * Positive exercise or chemical cardiac tolerance test
  * Patients currently under treatment for a medical condition requiring chronic use of steroids at a dose of prednisone >10 mg/day will be excluded.
  * Substance/alcohol abuse
  * Untreated proliferating diabetic retinopathy
  * PPD conversion or positive PPD without INH if suspicious TB by chest X-ray or symptoms
  * No primary care physician or primary care physician less than 6 months
  * Smoking in the last 6 months
  * Abnormal CBC / Hemoglobin < 10 g/dL
  * Microalbuminuria > 300 mg/24 hrs
  * Untreated hyperlipidemia - TC > 200 mg/dL, TGC > 200 mg/dL, LDL > 130 mg/dL
  * Untreated hyponatremia, hypokalemia, hypercalcemia, hypocalcemia
  * Iodine contrast allergy
  * PSA > 4 ng/mL
  * PRA > 20%
  * Active peptic ulcer disease/gallstones/hemangioma
  * Abnormal mammogram.
  * Patient receives any of the prohibited medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Restoration of sustained euglycemia without exogenous insulin or with reduced insulin dosage in patients who underwent pancreatic islet cell after kidney transplantation | 24 months
  Categorical variables will be analyzed using McNemar's test. Continuous data will be analyzed using repeated measures analysis of variance and Friedman's test when the normality assumption is violated. Follow-up pairwise comparisons will be performed using the Bonferroni multiple comparisons procedure at the 0.05 level of significance. Kaplan Meier estimates for patient and graft survival will be used.

SECONDARY OUTCOMES:
To assess incidence of hypoglycemic episodes | 24 months
To monitor insulin requirements in patients who did not achieve insulin independence | 24 months
To assess total islet mass needed to achieve sustained euglycemia with or without exogenous insulin. | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States